CLINICAL TRIAL: NCT04300530
Title: The Use of a Novel Monocyte Distribution Width (MDW) Biomarker of Infection in Hospital Practice
Brief Title: Monocyte Distribution Width (MDW) in Hospital Practice
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: St George's, University of London (Other)
Responsible Party: Sponsor
Other Study IDs: 2019.0376
Record Dates: First submitted 2020-03-03; First posted 2020-03-09 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Sepsis; Infection
Keywords: Monocyte Distribution Width; Sepsis; Infection; Cross-sectional Study
MeSH Terms: conditions — Sepsis; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Infections are an important cause of mortality and morbidity worldwide. Infections vary greatly in severity and can be caused by viruses, bacteria, fungi or protozoa. The rapid assessment of a patient to determine whether they have an infection and whether to treat with antibiotics is essential.

Monocyte Distribution Width (MDW) is a (CE marked) new biomarker that has recently been studied in the emergency department (ED). This novel biomarker, which is currently available as a part of the panel of results from full blood count, holds the promise of reducing unnecessary antibiotic use and improving the outcome of patient's infections.

Sepsis (blood poisoning) is a life-threatening condition that affects millions of people worldwide. The chance of dying from sepsis increases if there is a delay in treatment with the right antibiotics, but also using antibiotics incorrectly might lead to antibiotic resistance, which is dangerous for patients in the long term, as treatments might no longer work for them.

An antibiotic is a substance produced naturally by microorganisms or synthetically by chemists in a laboratory. Antibiotics are capable of inhibiting the growth of or killing bacteria but are not effective against the viruses that cause many illnesses. The inappropriate use of antibiotics for these types of non-bacterial infections as well as the more frequent use of broad-spectrum antibiotics has caused the emergence of newer strains of bacteria that are resistant to many antibiotics.

Rapid diagnostics are essential to accurately identify cases of sepsis that require antibiotic therapy; particularly since clinical criteria alone is often insufficient to avoid misclassifying patients with sepsis who require antibiotics. However, the high costs of current laboratory markers, along with the variable level of evidence supporting their use in sepsis and respiratory infections means that these are not in routine use.

This study proposes to make use of data collected routinely at St. George's University Hospital to evaluate the accuracy of MDW as a marker for sepsis in adult patients admitted to the ED, as well as to explore its usefulness in supporting clinical decisions related to the discontinuation of antibiotic treatment in hospitalised adult patients. This observational study will not involve changes in patient management as all the data would be analysed retrospectively.

DETAILED DESCRIPTION:
This is an observational, cross-sectional (single-gate) study comparing the results of the index test (MDW) against different reference standards (operational definitions). One of these references identifies a situation when IV antibiotics need to start (i.e. sepsis diagnosis) and the other, a situation when they need to be discontinued (i.e. clinical improvement).

One reference standard will be Sepsis 3 definition and will be operationalised in ED using qSOFA ≥ 2. This is used in ED as a bedside score to identify patients with suspected sepsis.

As part of the exploratory objectives for this ED dataset, sepsis will be operationalised using other common scores (SOFA, NEWS2, REDS, and Simplified-MISSED scores), and also against the reference standard for confirming septicaemia (blood culture results).

The second reference standard will be expert clinical criteria. Antimicrobial stewardship groups and care team review antibiotic treatments for all inpatients at regular intervals. Decisions on whether discontinuation (due to clinical improvement) is indicated is ultimately based on clinical criteria.

As part of the exploratory objectives for the dataset of in-patients, sepsis will be operationalised using the results of blood cultures. Also, different subpopulations will be described on the basis of MDW levels:

* Hospitalised patients admitted through ED but not in the sepsis pathway.
* Hospital Acquired Infections (HAI), surgical operations, and IV antibiotic treatment modification due to lack of clinical improvement and/or antibiotic resistance.
* Non-bacterial causes of septic syndrome (i.e. surgical tissue injury, myocardial infraction, pancreatitis, pulmonary-thromboembolism, influenza, RSV, autoimmune and neoplastic processes).

ELIGIBILITY:
Inclusion Criteria:

* Adults (aged ≥18 years).
* Patients who had at least one FBC requested between 01 January 2020 and 31 December 2020

Exclusion Criteria:

* Children and adolescents (< 18 years).
* Patients without a FBC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Coprimary objective 1: Admitted in ED for suspected sepsis between 01 January 2020 and 31 December 2020.
  Coprimary objective 2: Admitted to SGHFT wards for any reason between 01 January 2020 and 31 December 2020.
Sampling Method: Non-Probability Sample
Enrollment: 3098 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and Specificity of MDW to identify sepsis in adults presenting to the ED. | 1 day At ED admission
  Sensitivity and Specificity of MDW to identify sepsis in adults presenting to the ED against the reference clinical score, i.e. Sepsis 3 definition (operationalization of this definition in the ED is through qSOFA score).
Sensitivity and Specificity of MDW to predict clinical decisions related to IV antibiotic discontinuation in hospitalised adult patients. | 1 day At antibiotic discontinuation
  Sensitivity and Specificity of MDW to predict clinical decisions related to IV antibiotic discontinuation in hospitalised adult patients, against the current reference (clinical criteria). This will be measured when antibiotic treatment is assessed for discontinuation by direct care clinicians and stewardship team (the last full blood count at time of assessment will be used to obtain MDW values).

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - St. George's University Hospitals Foundation Trust, London
  - St. Georges Hospital Foundation Trust, London